CLINICAL TRIAL: NCT03389386
Title: Serum Catestatin Expression and Cardiometabolic Parameters in Patients With Congestive Heart Failure
Acronym: CATSTAT-HF
Status: Completed | Type: Observational
Sponsor: Josko Bozic (Other)
Collaborators: University of Split, School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Josko Bozic, Assistant Professor, University Hospital of Split
Organization: University Hospital of Split (Other)
Other Study IDs: 2181-147-01/06/M.S.-17-2
Record Dates: First submitted 2017-12-19; First posted 2018-01-03 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure，Congestive
Keywords: Congestive Heart Failure; Catestatin; Chromogranin A; Echocardiography; Biomarkers; Ventricular Dysfunction, Left; Comorbidity
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood obtained from the antecubital vein.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Congestive Heart Failure (NYHA II-IV): N=90
  Patients with a clinically documented diagnosis of congestive heart failure (CHF), as assessed per New York Heart Association (NYHA) functional classification will be prospectively and consecutively enrolled in this group. Patients will be of both sexes, enrolled in 1:1 ratio.
  All subjects in this group will undergo blood withdrawal for laboratory analysis, transthoracic echocardiography (TTE) examination and will be treated with the Standard-of-care treatment according to their current clinical condition at admission.
  Interventions: Diagnostic Test: Blood withdrawal for laboratory analysis; Other: Standard-of-care treatment; Diagnostic Test: Transthoracic echocardiography (TTE)
- Healthy Control Group: N=30
  Healthy volunteers (both sexes, enrolled in 1:1 ratio) with a negative history of cardiovascular diseases will be enrolled in this group that will serve as a study control.
  All subjects in this group will undergo blood withdrawal for laboratory analysis and transthoracic echocardiography (TTE) examination.
  Interventions: Diagnostic Test: Blood withdrawal for laboratory analysis; Diagnostic Test: Transthoracic echocardiography (TTE)

INTERVENTIONS:
Diagnostic Test: Blood withdrawal for laboratory analysis — Participants in this study will have their peripheral blood sampled from the cubital vein and the total volume withdrawn for the purposes of this study will be no more than 22 mL per person.
  Parameters of interest in the laboratory analysis will include serum catestatin levels, NT-proBNP levels, hs-cTnI, parameters of inflammation and renal function as well as standard biochemistry and complete blood count (CBC) panels.
Other: Standard-of-care treatment — Patients diagnosed with chronic heart failure will receive optimal standards of care in terms of pharmacologic management, according to their current clinical condition.
  Groups: Congestive Heart Failure (NYHA II-IV)
Diagnostic Test: Transthoracic echocardiography (TTE) — Participants from both groups will undergo transthoracic echocardiography examination that will measure established hemodynamic parameters of systolic and diastolic cardiac function as well as parameters of LV and RV strain in the selected subset of patients.

SUMMARY:
The congestive heart failure (HF) is a condition associated with substantial morbidity, mortality, and high healthcare expenditures. From the pathophysiological standpoint, several mechanisms contribute to the progression and dysfunction of the failing heart such as an increased hemodynamic overload, impaired myocyte calcium cycling, upregulated apoptotic activity, deficient or increased production of extracellular matrix, genetic predilections and, finally, excessive neurohumoral stimulation. The vasoactive neurohumoral systems such as sympathetic nervous system, renin-angiotensin-aldosterone system (RAAS) and arginine vasopressin (AVP) system all play a role in maintaining volume and circulatory homeostasis in the situation of impaired cardiac output.

Catestatin (CST), on another hand, is a novel endogenous peptide cleaved from chromogranin A (CgA) that is involved in the regulation of cardiac function and arterial blood pressure. The role of this peptide is to elicit potent catecholamine release-inhibitory activity by acting at the level of the nicotinic acetylcholine receptors. Therefore, the main hypothesis of this study is that the observed serum CST levels will reflect the degree of neurohormonal activation in HF, showing a significant relationship with the degree of disease severity as measured by relevant functional classifications (such as NYHA class and/or similar). Secondly, investigators expect to detect correlation of catestatin serum levels with the established risk stratification scores in HF and with the echocardiographic parameters of the ventricular function, both in terms of systolic and diastolic cardiac function. Parameters of inflammation, NT-proBNP, hs-cTnI, renal function parameters, and basic hematologic/biochemistry indices from peripheral blood will also be obtained and analyzed for all study participants.

Furthermore, according to the latest European Society of Cardiology (ESC) guidelines for the diagnosis and treatment of acute and chronic HF, participants with established congestive HF and the whole spectrum of left ventricular ejection fractions ranging from <40% to ≥50% will be included in the study.

Finally, all echocardiographic and laboratory parameters obtained from peripheral blood will be recorded and compared with respective healthy and matched control participants while participants diagnosed with HF will additionally be analyzed for potential differences between subgroups of interest.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women, 35-90 years of age
* Patients with clinically documented diagnosis of congestive heart failure (CHF) according to New York Heart Association (NYHA) functional classification (II-IV)

Exclusion Criteria:

* Age criteria:

  * Persons below legal age (<18 years)
  * Adults younger than 35 years of age
  * Adults older than 90 years of age
* Participants with following conditions:

  * Diabetes mellitus type I
  * Documented or newly-established severe valvular or pericardial disease
  * Infiltrative or hypertrophic cardiomyopathy
  * Primary pulmonary disease or cor pulmonale
  * Active malignant disease and/or active infectious disease
  * Significant systemic autoimmune disease
  * A positive history of excessive alcohol, drug, narcotics, and sedative consumption
  * Significant psychiatric or neurologic condition
  * Immunocompromised patients or patients that are under immunosuppressive treatment
  * Significant liver or renal insufficiency (primary renal or hepatic disease)
  * Hemorrhagic diathesis or significant coagulopathy
  * Positive recent history of cancer chemotherapeutic drug use
  * A positive history of acute coronary syndrome or stroke within 3 months prior to study enrollment

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the Congestive Heart Failure group will be consecutively enrolled from the pool of patients that will present with signs and symptoms of heart failure at Internal Medicine Emergency Department (ED) of the University Hospital of Split and will be subsequently admitted and hospitalized with working diagnosis of decompensated heart failure (I50.0). Patients that meet eligibility criteria and do not fulfill any of the excluding criteria will be further included in the study.
  Participants in the Healthy Control group will be enrolled from the sample of healthy residents of Split or nearby communities that meet the eligibility criteria for the study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Catestatin levels in blood serum | 3 months
  The goal is to determine and compare serum catestatin levels in patients with congestive heart failure, stratified by the left ventricular ejection fraction (LVEF) in three groups: reduced, mid-range, and preserved ejection fraction (HFrEF, HFmrEF, HFpEF). Furthermore, catestatin plasma levels will be compared between patients with congestive heart failure and healthy volunteers.

SECONDARY OUTCOMES:
Relationship of serum catestatin levels with the echocardiographic parameters of cardiac function | 3 months
  The potential relationship of catestatin serum levels with established parameters of systolic and diastolic cardiac function, as assessed by transthoracic echocardiography among patients with congestive heart failure will be examined.
Relationship of serum catestatin levels with the selected laboratory indices | 3 months
  The potential relationship of catestatin serum levels with the NT-proBNP, inflammatory biomarkers and standard hematologic/biochemical indices will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Josko Bozic, MD, PhD, Principal Investigator — Department of Pathophysiology, University of Split School of Medicine
Locations (1):
- University Hospital of Split, Split, Split-Dalmatia County, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borovac JA, Glavas D, Susilovic Grabovac Z, Supe Domic D, Stanisic L, D'Amario D, Kwok CS, Bozic J. Circulating sST2 and catestatin levels in patients with acute worsening of heart failure: a report from the CATSTAT-HF study. ESC Heart Fail. 2020 Oct;7(5):2818-2828. doi: 10.1002/ehf2.12882. Epub 2020 Jul 18. PMID 32681700
- [Derived] Borovac JA, Glavas D, Susilovic Grabovac Z, Supe Domic D, Stanisic L, D'Amario D, Duplancic D, Bozic J. Right Ventricular Free Wall Strain and Congestive Hepatopathy in Patients with Acute Worsening of Chronic Heart Failure: A CATSTAT-HF Echo Substudy. J Clin Med. 2020 May 2;9(5):1317. doi: 10.3390/jcm9051317. PMID 32370248
- [Derived] Borovac JA, Glavas D, Susilovic Grabovac Z, Supe Domic D, D'Amario D, Bozic J. Catestatin in Acutely Decompensated Heart Failure Patients: Insights from the CATSTAT-HF Study. J Clin Med. 2019 Jul 30;8(8):1132. doi: 10.3390/jcm8081132. PMID 31366074

DOCUMENTS (2):
  • Study Protocol (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03389386/Prot_004.pdf
  • Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03389386/SAP_005.pdf